CLINICAL TRIAL: NCT05877898
Title: ReCLaiMeD: Using Community Healthcare Workers to Improve Blood Pressure Control Among Food Insecure Hypertensive Adults: Aim 2
Brief Title: Improving Blood Pressure Control Among Food Insecure Hypertensive Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB202300592; UL1TR001427 (NIH)
Record Dates: First submitted 2023-05-17; First posted 2023-05-26 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-06

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No strategy (No Intervention): Individuals assigned to this arm with receive a publicly available color copy of the NIH's Healthy Blood Pressure for Healthy Hearts: Small Steps to Take Control Flyer available
- Community health worker provided education (Experimental): Participants will be invited to meet with the CHW to learn about eating healthier to reduce blood pressure and enhance quantity and quality of life. The CHW will register individuals for SNAP benefits and educate them on how to use their benefits locally. As other resources exist, including food pantries, food distribution events, and Fresh Access Bucks (a federal program to double SNAP if spent on local produce at eligible farmers markets), the CHW will provide information on these services. The CHW will also provide a brief motivational educational session about eating healthier to reduce BP and enhance quality and quantity of life. The CHW will meet once for up to one hour with each participant.
  Interventions: Behavioral: CHW Education
- Community health worker provided education and Navigation (Experimental): Participants will be invited to complete all the CHW education arm material and be offered a menu of optional services for personalization including: (1) transportation to the grocery store (weekly for 4 weeks), (2) culturally adapted hypertension-tailored cooking recipes, (3) a virtual cooking class with food delivered to their door led by community partner, (4) access to UF IFAS's online library of healthy food cooking videos, and (5) in-store education on food labels, grocery shopping, and food resource management skills through the Cooking Matters at the Store curricula.
  Interventions: Behavioral: CHW Education and Navigation

INTERVENTIONS:
Behavioral: CHW Education — Participants will be invited to meet with the CHW to learn about eating healthier to reduce blood pressure and enhance quantity and quality of life.
  Arms: Community health worker provided education
Behavioral: CHW Education and Navigation — Participants will be invited to complete all the CHW education arm material and be offered a menu of optional services for personalization including: (1) transportation to the grocery store (weekly for 4 weeks), (2) culturally adapted hypertension-tailored cooking recipes, (3) a virtual cooking class with food delivered to their door led by community partner, (4) access to UF IFAS's online library of healthy food cooking videos, and (5) in-store education on food labels, grocery shopping, and food resource management skills through the Cooking Matters at the Store curricula.
  Arms: Community health worker provided education and Navigation

SUMMARY:
The overall objective of this project is to assess the feasibility, acceptability, and appropriateness of adapted community health worker (CHW)-led implementation strategies designed to improve intake of fruits and vegetables and reduce BP among patients with hypertension experience food insecurity.

DETAILED DESCRIPTION:
We will recruit community members at food distribution events. Community members who have self-reported diagnosed hypertension, BP between 130 to 179 mm Hg systolic and 80 to 119 mm Hg diastolic, experience food insecurity (defined by the 10-question US Adult Food Security Survey Module), live in 32609, 32601, or 32641, are eligible for SNAP, are between 18 and 69 years old, and did not participate in our developmental focus groups are eligible for this study. Participants, will be invited to complete the baseline data collection, randomly assigned to a study group, and receive instructions on the next steps. The baseline data collection includes a brief behavior survey and baseline biometrics.

After the completion of the baseline data, participants will randomly be assigned to one of the three arms: (1) no strategy (n=25 participants), (2) Community Health Worker (CHW) education (n=25 participants), (3) CHW Education and Navigation (n=25 participants). Each participant will be in the study for the following 4 weeks.

The implementation strategies will be conducted by a trained and certified CHW from within the East Gainesville community. The participants assigned to no strategy will be provided a color copy of the NIH's Healthy Blood Pressure for Healthy Hearts: Small Steps to Take Control Flyer. The CHW Education arm participants will be invited to meet with the CHW to learn about eating healthier to reduce blood pressure and enhance quantity and quality of life. The CHW Education and Navigation arm participants will be invited to complete all the CHW education arm material and be offered a menu of optional services for personalization including: (1) transportation to the grocery store (weekly for 4 weeks), (2) culturally adapted hypertension-tailored cooking recipes, (3) a virtual cooking class with food delivered to their door led by community partnerr, (4) access to UF IFAS's online library of healthy food cooking videos, and (5) in-store education on food labels, grocery shopping, and food resource management skills through the Cooking Matters at the Store curricula.

We will produce descriptive statistics of baseline characteristics for study participants in each arm and test for balanced randomization. We will perform regression analyses, ANOVA estimations, and non-parametric statistical tests for pre-post differences in BP and carotenoid levels within and between treatment arms. Assuming a baseline systolic mean of 140 mmHg, standard deviation of 10, 25 participants/arm, and alpha 0.05, we will have 82% power to detect a 8 mmHg difference in both active arms vs. control, similar to prior dietary studies (≥71% power if one arm achieves only 4 mmHg difference). Average scores of ≥3 on the 0-5 scale for AIM, FIM, and IAM will indicate success.

ELIGIBILITY:
Inclusion Criteria:

* self-reported diagnosed hypertension
* BP between 130 to 179 mm Hg systolic and 80 to 119 mm Hg diastolic
* experience food insecurity
* live in 32609, 32601, or 32641 zip codes
* eligible for SNAP

Exclusion Criteria:

* Participated in a focus group to develop the intervention

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-05-27 (Actual); Study Completion 2025-05-27 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 4 weeks
  Change in measure of participant systolic and diastolic blood pressure
carotenoid levels | 4 weeks
  Change in carotenoid levels as measured by the Veggie Meter

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Staras, PhD, Principal Investigator — University of Florida; Carla Fisher, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-02-21): https://cdn.clinicaltrials.gov/large-docs/98/NCT05877898/ICF_000.pdf